CLINICAL TRIAL: NCT00312585
Title: A Randomized Controlled Trial of Acupuncture to Prevent Postdates Pregnancy
Brief Title: Acupuncture for the Prevention of Postdates Pregnancy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Responsible Party: Remy Coeytaux, MD, University of North Carolina at Chapel Hill
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: G0418
Record Dates: First submitted 2006-04-06; First posted 2006-04-10 (Estimated); Last update posted 2016-04-07 (Estimated); Status verified 2011-05

CONDITIONS: Pregnancy
Keywords: pregnancy; acupuncture
MeSH Terms: interventions — Acupuncture Therapy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Acupuncture (Experimental)
  Interventions: Procedure: Acupuncture
- Sham Acupuncture (Sham Comparator)
  Interventions: Procedure: Sham comparator
- Usual care only (No Intervention)

INTERVENTIONS:
Procedure: Acupuncture
  Arms: Acupuncture
Procedure: Sham comparator
  Arms: Sham Acupuncture

SUMMARY:
The purpose of this study is to assess if acupuncture can shorten the time to delivery for women who are experiencing their first, full-term pregnancy.

DETAILED DESCRIPTION:
There are certain medical conditions that can complicate pregnancies after 40 weeks gestation. However, it is not always safe or easy to put these women into labor. Acupuncture has been used in Asia for hundreds of years to induce contractions and begin the labor process. Acupuncture is not typically used in the United States to induce labor, however. The purpose of this study is to determine whether a series of up to five acupuncture treatments can prevent postdates pregnancy.

ELIGIBILITY:
Inclusion Criteria:

* first, full-term pregnancy
* 38-41 weeks gestation
* English or Spanish speaking
* Bishop score of 7 or less

Exclusion Criteria:

* uncertain pregnancy dating
* transportation difficulties
* previous inability to tolerate acupuncture
* age less than 18

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 89 (Actual)
Dates: Start 2005-02; Primary Completion 2007-03 (Actual); Study Completion 2007-03 (Actual)

PRIMARY OUTCOMES:
prevention of inpatient induction of labor

SECONDARY OUTCOMES:
rate of cesarean delivery
rates of chorioamnionitis
length of maternal hospital stay
rates of assisted delivery
neonatal outcomes

CONTACTS AND LOCATIONS:
Overall Officials: Teresa Harper, MD, Principal Investigator — UNC-Chapel Hill Department of Ob/Gyn
Locations (1):
- UNC-Chapel Hill Family Medicine Center, Chapel Hill, North Carolina, United States

REFERENCES:
- [Result] Harper TC, Coeytaux RR, Chen W, Campbell K, Kaufman JS, Moise KJ, Thorp JM. A randomized controlled trial of acupuncture for initiation of labor in nulliparous women. J Matern Fetal Neonatal Med. 2006 Aug;19(8):465-70. doi: 10.1080/14767050600730740. PMID 16966110